CLINICAL TRIAL: NCT01029093
Title: Effects of Sensory and Motor Deprivation on Brain Plasticity After Injury and Immobilisation of Right Upper Extremity
Brief Title: Effects of Sensory and Motor Deprivation on Brain Plasticity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Collaborators: Jaencke (Unknown)
Responsible Party: Hans-Peter Simmen MD Professor and Chair Division of Trauma Surgery and Prof. Dr. rer. nat. Lutz Jäncke, Chief of Division Neuropsycholoy, Institute Psychology, University Zurich, Division of Trauma Surgery and Institute of Psychology, Division Neuropsycholgy, University Zurich
Other Study IDs: Ref-Nr: StV 13-2009
Record Dates: First submitted 2009-11-25; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Injury of the Right Upper Extremity
Keywords: extremity with immobilisation; brain platicity; deprivation; MRI
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: no intervention, MRI and motor skill test — Two MR Investigations at two different times
  Other Names: MRI; motor skill test

SUMMARY:
Investigation of changes in gray and white matter during immoblisation after injury of the right upper extremity via two MR Investigations of the brain at two different times.

DETAILED DESCRIPTION:
Investigation of changes in gray and white matter during immoblisation after injury of the right upper extremity via two MR Investigations of the brain at two different times. Immobilisation at least 12 days. Time between the 2 investigations: 12-14 d.

ELIGIBILITY:
Inclusion criteria:

* Right handed
* Injury of right upper extremity where immobilisation is needed

Exclusion criteria:

* TBI, neurological or psychatric deseases
* Other cerebral deseases
* Standard MRI Exclusion criterias such as pacemaker, epilepsia etc

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with injury of right upper extremity
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Devision of Traum, Zurich, Switzerland